CLINICAL TRIAL: NCT04031118
Title: Corneal Oxygen Uptake With Apioc Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lentechs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Device Feasibility
Other Study IDs: Len-003
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Contact Lens-Induced Corneal Disorder of Both Eyes (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Apioc Contact Lens — Measurement of corneal oxygen uptake with contact lens wear.

SUMMARY:
The purpose of this research is to determine if a new investigational contact lens shape allows the eye to get more oxygen.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent.
2. Appear willing and able to adhere to instructions set forth in the protocol.
3. Be between the ages of 18 and 45.
4. Be an experienced contact lens wearer.
5. Be an eyecare clinician or clinician-in-training.
6. Flat and steep keratometry readings within 40 to 50D.
7. Clear, healthy corneas with no irregular astigmatism.
8. Normal, healthy conjunctiva in both eyes.
9. Be able to provide corneal topography measurements.
10. Be able to provide manifest refraction measurements.

Exclusion Criteria:

1. Irregular corneal astigmatism.
2. Use of topical or systemic antihistamines within the previous week.
3. Use of topical ophthalmic drops within the previous two days.
4. History of corneal surgery.
5. Currently pregnant or lactating.
6. Systemic disease that would interfere with contact lens wear.
7. Previous diagnosis of dry eye syndrome.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Corneal Oxygen Uptake Rate | up to 45 seconds
  uptake of oxygen by human cornea in vivo

CONTACTS AND LOCATIONS:
Locations (1):
- Rev1 Ventures, Columbus, Ohio, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04031118/Prot_SAP_000.pdf